CLINICAL TRIAL: NCT05172648
Title: Effect of Small-volume Oral Spray in the After Anesthesia Recovery Room for Thirst Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202104124RINC
Record Dates: First submitted 2021-11-21; First posted 2021-12-29 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2021-11

CONDITIONS: Anesthesia and Thirst
Keywords: thirst and oral spray and after anesthesia and recovery room

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Pour sterile distilled water into a 30ml small-capacity spray bottle and spray 4 times at the patient's mouth. They are on the tongue and under the tongue, the left side and the right side of the mouth. The same spray bottle is used by the same person. Consistent dosage and strength
  Interventions: Other: oral spry
- contrast group (Other): Moisten the mouth with sterile distilled water with an oral cotton swab.
  Interventions: Other: Cotton swab

INTERVENTIONS:
Other: oral spry — Pour sterile distilled water into a 30ml small-capacity spray bottle and spray 4 times at the patient's mouth. They are on the tongue and under the tongue, the left side and the right side of the mouth. The same spray bottle is used by the same person. Consistent dosage and strength.
  Arms: control group
Other: Cotton swab — Moisten the mouth with sterile distilled water with an oral cotton swab.
  Arms: contrast group

SUMMARY:
Currently, there are limited studies performed on the treatment of perioperative thirst and the methods provided by literature possess a risk of choking. In addition, there is no good treatment nor relevant research in the area of perioperative thirst in Taiwan. As a result, this study aims to use a visual analogue scale (VAS) as the assessment tool to show that oral spray can significantly ease the thirst-related discomfort for patients recovering from anesthesia, thereby reducing the frequency of painkiller use. This would result in lower labor and material costs, achieving the effect of improved perioperative care quality and cost reduction. It is hoped that in the future, the study can be applied in practice and academic studies to reduce perioperative thirst for patients. Using patients with perioperative thirst in the recovery room as the subject, this study planned to have research personnel or part-timers collect data from a total of 200 patients. Statistical analysis would be performed for data collected from the recovery room.

DETAILED DESCRIPTION:
Research design and research subjects use surveymonkey's sample number calculator to set the total number of patients in the year before inclusion and exclusion as the mother population: 5600, the verification power is set to 0.8, the effect is set to 5%, and the estimated sample number needs to be at least 160 patient. The admission process is shown in Figure 1. After the patient reports in the operation registration area, the admission officer randomly selects at least 3 non-head and neck surgery patients every day (see the inclusion and exclusion conditions for details), and gives written and verbal explanations, and obtains informed consent and Signing the consent form, deducting the number of samples lost (for example, the lips are broken due to the intraoperative intubation process or the VAS thirst assessment form score is less than 4 points), and it is estimated that a total of 300 patients will be enrolled. After the patients enter the recovery room, those eligible for inclusion are divided into the control group, the oral spray group and the control group, the oral spray group and the control group, after the sample is lost, it is expected that each group will receive 100 patients. Inclusion conditions: VAS thirst assessment form score ≥ 4 points, age 20-75 years old, anesthesia risk assessment grade ASA: I~III, conscious (GCS: 15 points), Muscle power ≥ 4 points, anesthesia recovery score Aldrate score ≥8 points, informed consent. Excluded conditions: Those who have undergone head and neck surgery this time or have a history of head and neck surgery, have diabetes, hyperthyroidism, a history of heart failure, are younger than 20 years old or older than 75 years old, or have broken oral mucosa or lips.

Research tools: 30ml small-capacity spray bottle, oral cotton swab, sterile distilled water, VAS thirst visual assessment form.

Steps of the study: After entering the recovery room, the patients who meet the criteria for inclusion are divided into the control group, the oral spray group (singular) and the control group, the cotton swab moisturizing the mouth group using random random number generators (minimum 1, maximum 10) (Double number), after the patient wakes up (Aldrate score ≥ 8 points), VAS thirst visual assessment scale score ≥ 4 points, immediately intervene. The control group poured sterile distilled water into a 30ml small-capacity spray bottle and sprayed it on the patient's mouth 4 times, respectively on the oral tongue and under the tongue, the left side and the right side of the mouth. The dose and intensity of the spray were the same; the control group used an oral cotton swab to moisten the oral cavity with sterile distilled water. Before the first intervention and before being transferred out of the recovery room, the VAS Thirst Assessment Form was used to score a total of 2 assessments. In addition, retrospective statistics.

ELIGIBILITY:
Inclusion Criteria:

1. VAS thirst assessment form score ≥ 4 points
2. Age 20-75 years old
3. Anesthesia risk assessment grade Amersican Society of Anesthesiologists: I~III:The first level (ASAⅠ)-healthy people, except for surgical corrections, without any systemic disease patients, such as patients with simple appendicitis (pre- and post-operative mortality rate 0.06~0.08%); Level 2 (ASAⅡ)-Patients with mild systemic disease but no functional impairment, such as those over 70 years old without any disease, or a small cold, HTN or DM but well-controlled diseases (pre- and post-operative mortality 0.27~0.4%); Level III (ASAⅢ)-Moderate to severe systemic disease and cause partial dysfunction, such as HTN or DM but not well controlled, or have cardiovascular complications (stroke, myocardial infarction, angina, etc.) (The mortality rate before and after surgery is 1.8~4.3%).
4. Conscious (GCS: 15 points).
5. Muscle power ≥ 4 points.
6. Anesthesia recovery score Aldrate score ≥8 points: Consciousness: Fully awake, in full contact; Mobility: Able to move 2 extremities on command; Breathing: Able to breathe deeply and cough freely; Circulation: BP ±20-49% of pre-anesthetic level; Skin color: Normal.
7. Informed consent.

Excluded Criteria:

1. Those who underwent head and neck surgery this time or had a history of head and neck surgery: Acoustic immittance testing, Acoustic voice assessment, Aerodynamic voice assessment, Airway reconstruction, Auditory brainstem implant, Auditory evoked potential test, Aural rehabilitation, Balloon sinuplasty, Blepharoplasty, Botox injections, Bronchoscopy, Brow lift, Canalith repositioning procedure, Chemical peel, Cleft lip repair, Cleft palate repair, CO-2 laser treatment, Cochlear implants, Computerized dynamic posturography, Cosmetic surgery, Custom ear protector fitting, Dental implant surgery, Electroacoustic assessments of hearing aids, Electromyography (EMG), Electronystagmography, Endoscopic sinus surgery, Esophagoscopy, Face-lift, Facial fillers for wrinkles, Facial fracture repair, Facial nerve rehabilitation, Facial reconstruction, Facial rejuvenation, Fat grafting, Flexible endoscopic evaluation of swallowing with sensory, testing (FEESST), Hearing aid fitting, Hearing conservation services, Hearing implant surgery, Hearing monitoring services, Hearing test, Hearing test for children, Infant hearing screening, KTP laser treatment, Laryngeal reinnervation, Laryngoscopy, Laryngotracheal reconstruction, Larynx transplant, Laser resurfacing, Lip surgery, Mastoidectomy, Maxillomandibular advancement surgery, Microlaryngoscopy, Microvascular reconstruction, Middle ear reconstruction, Minimally invasive surgery, Nasal septal reconstruction, Nasal valve repair, Neck lift, Newborn hearing screening, Nose reconstruction, Otoacoustic emissions (OEA) test, Otological microsurgery, Otoplasty, Parathyroidectomy, Parotid gland surgery, Parotidectomy, Pharyngeal manometry, Professional voice evaluation, Rhinoplasty, Robotic surgery, Rotary-chair testing, Scar revision, Septoplasty, Singing voice evaluation, Sinus surgery, Skin cancer reconstruction, Speech-language pathology evaluation, Stapedectomy, Stroboscopy, Swallowing exercises, Swim mold fitting, Thyroid surgery, Thyroidectomy, Thyroplasty, Tinnitus assessment, Tonsillectomy, Trachea transplant, Tracheostomy, Transnasal esophagoscopy, Transnasal pituitary surgery, Transoral laser microsurgery, Transoral robotic surgery, Turbinate surgery, Ultrasound-guided fine-needle aspiration, Ultrasound-guided surgery, Upper airway stimulation therapy (Inspire device), Uvulopalatopharyngoplasty (UPPP), Vestibular rehabilitation, Vestibular testing, Videofluoroscopic swallowing study, Video laryngoscopy, Vocal cord injection, Voice therapy.
2. A history of Diabetes.
3. A history of Hyperthyroidism.
4. A history of heart failure
5. Younger than 20 years old or older than 75 years old.
6. Damaged oral mucosa or lips.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale of Thirst Assessment( minimum values: 0, maximum values: 10) | 1hour
  Before the first intervention and before being transferred out of the recovery room, use the Visual Analogue Scale of Thirst Assessment( minimum values: 0, maximum values: 10) Form to score a total of 2 times.

SECONDARY OUTCOMES:
Number of painkillers used | 1hour
  In addition, retrospective statistics were used to determine whether there was a difference in the number of thirst interventions and the number of painkillers used between the two groups of patients.

CONTACTS AND LOCATIONS:
Overall Officials: ChingWen Cheng, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Test2, Taiwan